CLINICAL TRIAL: NCT03028142
Title: The Effects of RPL554 in Addition to Tiotropium in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RPL554-CO-202
Record Dates: First submitted 2017-01-03; First posted 2017-01-23 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-01

CONDITIONS: Chronic Obstructive Pulmonary Disease Moderate
MeSH Terms: interventions — ensifentrine; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lower Dose Nebulised Treatment (Experimental): 1.5 mg nebulised RPL554 twice daily plus 10 mcg tiotropium DPI once daily for 3 days
  Interventions: Drug: 1.5 mg RPL554 plus tiotropium
- Higher Dose Nebulised Treatment (Experimental): 6 mg nebulised RPL554 twice daily plus 10 mcg tiotropium DPI once daily for 3 days
  Interventions: Drug: 6 mg RPL554 plus tiotropium
- Placebo (Placebo Comparator): Nebulised RPL554 matched placebo twice daily plus 10 mcg tiotropium DPI once daily for 3 days
  Interventions: Drug: Placebo plus tiotropium

INTERVENTIONS:
Drug: 1.5 mg RPL554 plus tiotropium
  Arms: Lower Dose Nebulised Treatment
Drug: 6 mg RPL554 plus tiotropium
  Arms: Higher Dose Nebulised Treatment
Drug: Placebo plus tiotropium
  Arms: Placebo

SUMMARY:
This is a phase II, randomised, double blind, placebo controlled, complete block, three way crossover study to investigate treatment with nebulised RPL554 and tiotropium together in patients with moderate to severe chronic obstructive pulmonary disease (COPD). The purpose of this study is to assess the bronchodilator effect (opening of the airways) of RPL554 when used in combination with a long acting anti-muscarinic receptor antagonist (tiotropium) whilst dosing the RPL554 to steady state blood levels. It is planned to randomise up to 30 patients to have 24 evaluable patients at one study centre. In each treatment period, patients will receive an open label dose of tiotropium from a dry power inhaler (DPI) followed immediately by a double blind dose of either RPL554 6mg, 1.5mg or placebo (depending on treatment sequence) from a nebuliser in the morning on Day 1, Day 2 and Day 3. The dose of RPL554 or placebo will be repeated in the evening on Day 1 and Day 2; there will not be an evening dose on Day 3.

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study.
2. Male or female aged between 40 and 75 years inclusive, at the time of informed consent.
3. If male: must agree to meet the following from the first dose up to 1 month after the last dose of study treatment:

   * Not donate sperm
   * Either: be sexually abstinent in accordance with a patient's usual and preferred lifestyle (but agree to abide by the contraception requirements below should their circumstances change) Or: use a condom with all sexual partners. If the partner is of childbearing potential the condom must be used with spermicide and a second highly effective form of contraception must also be used
4. If female: either be:

   1. Of non-childbearing potential defined as being:

      * Either: post-menopausal (being spontaneously amenorrhoeic for at least 1 year with an appropriate clinical profile [e.g. age appropriate, history of vasomotor symptoms]
      * Or: permanently sterilised e.g. tubal occlusion, hysterectomy, bilateral oophorectomy, bilateral salpingectomy
   2. Of childbearing potential and agreeing to use a highly effective method of contraception until completion of the end of study visit.
5. Have a 12-lead ECG recording at screening and randomisation (pre-dose in Treatment Period 1) showing the following:

   * Heart rate between 45 and 90 beats per minute (bpm)
   * QT interval corrected for heart rate using Fridericia's formula (QTcF) ≤450 msec for males and ≤470 ms for females
   * QRS interval ≤120 msec
   * No clinically significant abnormalities (as judged by the Investigator) including morphology (e.g. left bundle branch block, atrio-ventricular nodal dysfunction, ST segment abnormalities)
6. Have a screening Holter report with a minimum of 18 hours recording that is able to be evaluated for rhythm analysis which shows no abnormality which indicates a significant impairment of patient safety or which may significantly impairs interpretation in the opinion of the Investigator including:

   * Significant arrhythmias including atrial flutter, atrial fibrillation, ventricular tachycardia
   * Any symptomatic arrhythmia (except isolated extra systoles)
   * Any sustained second or third degree heart block
7. Capable of complying with all study restrictions and procedures including ability to use the study nebuliser and HandiHaler® DPI correctly.
8. Body mass index (BMI) between 18 and 33 kg/m2 (inclusive) with a minimum weight of 45 kg.
9. COPD diagnosis: Patients with a diagnosis of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines (Celli and MacNee, 2004) with symptoms compatible with COPD for at least 1 year prior to screening.
10. Post-bronchodilator (four puffs of salbutamol) spirometry at screening:

    * Post-bronchodilator forced expiratory volume in 1 second (FEV1)/forced vital capacity (FVC) ratio of ≤0.70
    * Post-bronchodilator FEV1 ≥40 % and ≤80% of predicted normal
    * Demonstrates ≥150 mL increase from pre-bronchodilator FEV1
11. Clinically stable COPD in the 4 weeks prior to screening and randomisation (pre-dose in Treatment Period 1).
12. A chest X-ray (post-anterior) at screening, or in the 12 months prior to screening showing no abnormalities, which are both clinically significant and unrelated to COPD.
13. Meet the concomitant medication restrictions and be expected to do so for the rest of the study.
14. Smoking history of ≥10 pack years.
15. Capable of withdrawing from long acting bronchodilators for the duration of the study, and short acting bronchodilators for 8 hours prior to spirometry.

Exclusion Criteria:

1. A history of life-threatening COPD exacerbation including Intensive Care Unit admission and/or requiring intubation.
2. COPD exacerbation requiring oral steroids, or lower respiratory tract infection requiring antibiotics, in the 3 months prior to screening or randomisation (pre-dose in Treatment Period 1).
3. A history of one or more hospitalisations for COPD in the 12 months prior to screening or randomisation (pre-dose in Treatment Period 1).
4. Lactation (female patients only).
5. Positive urine or serum pregnancy test at screening, or a positive urine pregnancy test prior to randomisation (female patients of childbearing potential only).
6. Prior exposure to RPL554 or known hypersensitivity to RPL554 or its components.
7. Intolerance or hypersensitivity to tiotropium.
8. Evidence of cor pulmonale.
9. Other respiratory disorders: Patients with a current diagnosis of asthma, active tuberculosis, lung cancer, bronchiectasis, sarcoidosis, lung fibrosis, interstitial lung diseases, sleep apnoea, known alpha-1 antitrypsin deficiency or other active pulmonary diseases.
10. Previous lung resection or lung reduction surgery.
11. Use of oral COPD medications (e.g. oral steroids, theophylline and romifulast) in the 3 months prior to screening or randomisation (pre-dose in Treatment Period 1).
12. History of, or reason to believe, a patient has drug or alcohol abuse within the past 3 years.
13. Inability to perform technically acceptable spirometry or whole body plethysmography (at screening or randomisation [pre dose in Treatment Period 1])
14. Received an experimental drug within 30 days or five half lives, whichever is longer.
15. Patients with a history of chronic uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, haematological, urological, immunological, or ophthalmic diseases that the Investigator believes are clinically significant.
16. Documented cardiovascular disease: arrhythmias, angina, recent or suspected myocardial infarction, congestive heart failure, a history of unstable, or uncontrolled hypertension, or has been diagnosed with hypertension in the 3 months prior to screening or randomisation.
17. Concurrent use of non-cardioselective oral beta-blockers.
18. Has had major surgery, (requiring general anaesthesia) in the 6 weeks prior to screening or randomisation (pre-dose in Treatment Period 1), or will not have fully recovered from surgery, or planned surgery through the end of the study.
19. A disclosed history or one known to the Investigator, of significant non compliance in previous investigational studies or with prescribed medications.
20. Requires oxygen therapy, even on an occasional basis.
21. Clinically significant prostatic hyperplasia (judged by the Investigator) or bladder-neck obstruction or with narrow-angle glaucoma.
22. Any other reason that the Investigator considers makes the patient unsuitable to participate.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singh D, Abbott-Banner K, Bengtsson T, Newman K. The short-term bronchodilator effects of the dual phosphodiesterase 3 and 4 inhibitor RPL554 in COPD. Eur Respir J. 2018 Nov 1;52(5):1801074. doi: 10.1183/13993003.01074-2018. Print 2018 Nov. PMID 30166326

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 74 were screened.Main reasons for screen failure were reversibility criteria not met (21), withdrew consent (5) and unsuitable chronic obstructive pulmonary disorder (COPD) history (4). Patients had to discontinue long acting bronchodilators on the day before screening and short acting bronchodilators for 8 hours before all spirometry assessments
Groups:
- Placebo Then Low Dose RPL554 Then High Dose RPL554: Placebo twice daily plus 10 mcg tiotropium once daily for 3 days then 1.5 mg RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then 6 mg RPL554 twice daily plus 10 mcg tiotropium for 3 days, with a 7-21 day washout period between treatments
- Low Dose Dose RPL554 Then High Dose RPL554 Then Placebo: 1.5 mg RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then 6 mg RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then placebo twice daily plus 10 mcg tiotropium for 3 days, with a 7-21 day washout period between treatments
- High Dose RPL554 Then Placebo Then Low Dose RPL554: High dose RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then placebo twice daily plus 10 mcg tiotropium once daily for 3 days then 1.5 mg RPL554 twice daily plus 10 mcg tiotropium for 3 days, with a 7-21 day washout period between treatments
- High Dose RPL554 Then Low Dose RPL554 Then Placebo: High dose RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then 1.5 mg RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then placebo twice daily plus 10 mcg tiotropium for 3 days, with a 7-21 day washout period between treatments
- Low Dose RPL554 Then Placebo Then High Dose RPL554: Low dose RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then placebo twice daily plus 10 mcg tiotropium once daily for 3 days then 6 mg RPL554 twice daily plus 10 mcg tiotropium for 3 days, with a 7-21 day washout period between treatments
- Placebo Then High Dose RPL554 Then Low Dose RPL554: Placebo twice daily plus 10 mcg tiotropium once daily for 3 days then 6 mg RPL554 twice daily plus 10 mcg tiotropium once daily for 3 days then 1.5 mg RPL554 twice daily plus 10 mcg tiotropium for 3 days, with a 7-21 day washout period between treatments
Period: Overall Study
Arm/Group | Placebo Then Low Dose RPL554 Then High Dose RPL554 | Low Dose Dose RPL554 Then High Dose RPL554 Then Placebo | High Dose RPL554 Then Placebo Then Low Dose RPL554 | High Dose RPL554 Then Low Dose RPL554 Then Placebo | Low Dose RPL554 Then Placebo Then High Dose RPL554 | Placebo Then High Dose RPL554 Then Low Dose RPL554
Started | 5 | 5 | 6 | 4 | 6 | 4
Completed | 4 | 4 | 6 | 4 | 5 | 3
Not Completed | 1 | 1 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All patients who received at least one dose of study treatment
Groups:
- Overall: All patients before the start of the study treatment sequence
Arm/Group | Overall
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 64.5 [47 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Percentage of predicted FEV1 post-bronchodilator [Mean (Standard Deviation); unit: %] | 60.1 (9.73)

OUTCOME MEASURES:

1. Primary Outcome: Peak Forced Expired Volume in 1 Second (FEV1) on the Third Day of Dosing
Description: Peak forced expired volume in 1 second (FEV1) over 4 hours on the third day of dosing
Time Frame: Day 3
Population: All randomized patients with sufficient data collected after intake of study treatment to compute the pharmacodynamics parameters on at least two treatment periods.
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Lower Dose Nebulised Treatment: 1.5 mg nebulised RPL554 twice daily plus 10 mcg tiotropium dry powder inhaler (DPI) once daily for 3 days
  1.5 mg RPL554 plus tiotropium
- Higher Dose Nebulised Treatment: 6 mg nebulised RPL554 twice daily plus 10 mcg tiotropium DPI once daily for 3 days
  6 mg RPL554 plus tiotropium
- Placebo: Nebulised RPL554 matched placebo twice daily plus 10 mcg tiotropium DPI once daily for 3 days
  Placebo plus tiotropium
Arm/Group | Lower Dose Nebulised Treatment | Higher Dose Nebulised Treatment | Placebo
Number analyzed (Participants) | 28 | 27 | 27
Liters | 0.477 (0.1673) | 0.500 (0.2157) | 0.373 (0.1970)
Statistical Analysis 1: Comparison: Lower Dose Nebulised Treatment vs Placebo; Test type: Other; p = 0.0022, ANCOVA; LS Means ratio = 1.05, 95% CI 2-sided [1.02 to 1.09]
Statistical Analysis 2: Comparison: Higher Dose Nebulised Treatment vs Placebo; Test type: Other; p < 0.0001, ANCOVA; LS Means ratio = 1.09, 95% CI 2-sided [1.05 to 1.12]

2. Primary Outcome: Average FEV1 Over 12 Hours on the Third Day of Dosing
Description: Average FEV1 area under the curve (AUC) over 12 hours on the third day of dosing
Time Frame: Day 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters*hour
Groups:
- Lower Dose Nebulised Treatment: 1.5 mg nebulised RPL554 twice daily plus 10 mcg tiotropium DPI once daily for 3 days
  1.5 mg RPL554 plus tiotropium
Arm/Group | Lower Dose Nebulised Treatment | Higher Dose Nebulised Treatment | Placebo
Number analyzed (Participants) | 28 | 27 | 27
Liters*hour | 3.804 (1.8512) | 3.967 (2.2134) | 3.197 (2.2826)
Statistical Analysis 1: Comparison: Lower Dose Nebulised Treatment vs Placebo; Test type: Other; p = 0.0988, ANCOVA; LS Means ratio = 1.03, 95% CI 2-sided [0.99 to 1.06]
Statistical Analysis 2: Comparison: Higher Dose Nebulised Treatment vs Placebo; Test type: Other; p = 0.0009, ANCOVA; LS Means ratio = 1.06, 95% CI 2-sided [1.02 to 1.09]

3. Secondary Outcome: Peak FEV1 on Day 1
Description: Peak FEV1 over 4 hours on Day 1
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lower Dose Nebulised Treatment | Higher Dose Nebulised Treatment | Placebo
Number analyzed (Participants) | 28 | 27 | 27
Liters | 0.383 (0.1448) | 0.432 (0.1720) | 0.337 (0.1854)
Statistical Analysis 1: Comparison: Lower Dose Nebulised Treatment vs Placebo; Test type: Other; p = 0.2496, ANCOVA; LS Means ratio = 1.02, 95% CI 2-sided [0.98 to 1.06]
Statistical Analysis 2: Comparison: Higher Dose Nebulised Treatment vs Placebo; Test type: Other; p = 0.0039, ANCOVA; LS Means ratio = 1.06, 95% CI 2-sided [1.02 to 1.1]

4. Secondary Outcome: Average FEV1 Over 12 Hours on Day 1
Description: Average FEV1 AUC over 12 hours on Day 1
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: Liters*hour
Arm/Group | Lower Dose Nebulised Treatment | Higher Dose Nebulised Treatment | Placebo
Number analyzed (Participants) | 28 | 27 | 27
Liters*hour | 3.058 (1.4851) | 3.094 (1.9624) | 2.510 (1.9381)
Statistical Analysis 1: Comparison: Lower Dose Nebulised Treatment vs Placebo; Test type: Other; p = 0.1404, ANCOVA; LS Means ratio = 1.03, 95% CI 2-sided [0.99 to 1.06]
Statistical Analysis 2: Comparison: Higher Dose Nebulised Treatment vs Placebo; Test type: Other; p = 0.0228, ANCOVA; LS Means ratio = 1.04, 95% CI 2-sided [1.01 to 1.08]

ADVERSE EVENTS:
Time Frame: From informed consent until the end of the study.
Arm/Group | Lower Dose Nebulised Treatment | Higher Dose Nebulised Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 1/29 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 12/29 | 12/27 | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose Nebulised Treatment (N=29) | Higher Dose Nebulised Treatment (N=27) | Placebo (N=28)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Dose Nebulised Treatment (N=29) | Higher Dose Nebulised Treatment (N=27) | Placebo (N=28)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (3)
Headache (Nervous system disorders) | 2 (2) | 5 (8) | 3 (3)
Medical device site reaction (General disorders) | 4 (4) | 1 (1) | 4 (4)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 2 (3)
Catheter site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Larngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The employees of the Medicines Evaluation shall not be permitted to present at symposia, national or regional professional meetings, and to publish in journals, theses or dissertations, or otherwise of their own choosing, methods and results of the Clinical Trial subject to the publication policy described in the Protocol without prior written approval of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03028142/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT03028142/SAP_001.pdf